CLINICAL TRIAL: NCT06264622
Title: Dose Response Study of the Effects of a Daily Supplementation With a Black Garlic Extract, ABG+/GarlACE on Cardiovascular Disease Risk Factors in Subjects With Grade I Hypertension
Brief Title: ABG+/GarlACE Effects on Cardiovascular Risk Factors in Subjects With Grade I Hypertension
Acronym: GARDOSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Collaborators: Pharmactive Biotech Products S.L.U (Industry)
Responsible Party: Principal Investigator, José Serrano, Professor, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEIC-2996
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hypertension
Keywords: Grade I Hypertension
MeSH Terms: conditions — Hypertension | interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): 250 mg/day of Garlic Extract
  Interventions: Dietary Supplement: Low dose
- High Dose (Experimental): 600 mg/day of Garlic Extract
  Interventions: Dietary Supplement: High dose
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Low dose — 2 tablets per day during the morning for 12 weeks.
  Arms: Low Dose
Dietary Supplement: High dose — 2 tablets per day during the morning for 12 weeks.
  Arms: High Dose
Dietary Supplement: Placebo — 2 tablets per day during the morning for 12 weeks.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the dose response effect on cardiovascular disease risk factors of a Black Garlic Extract in subjects with Grade I Hypertension. The main questions it aims to answer are:

* If the reduction in blood pressure (systolic and diastolic) is in a dose-response manner
* If the changes in lipid profile are in a dose-response manner

Participants will be randomly assign to a low dose (250 mg/day), high dose (600 mg/day) or placebo of a standardized Garlic Extract (ABG+/GarlACE) during 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Men and women with Grade I Hypertension (systolic blood pressure between 130 and 139 mmHg; and diastolic blood pressure between 80 to 89 mmHg) without taking any antihypertensive drug

Exclusion Criteria:

* Acute or chronic kidney disease including dyslipidemia due to nephrotic syndrome.- -
* Hypothyroidism
* Having previously suffered a myocardial infarction or stroke
* Pharmacological treatment with insulin, sulfonylureas, protease inhibitors
* Chronic gastrointestinal disease
* Pregnancy or intention to become pregnant during the study period.
* Breastfeeding
* Allergy or intolerance to garlic
* High alcohol consumption (>14 units per week)
* Smokers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-26 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Pre-treatment and 12 weeks post-treatment
  Upper arm blood pressure (Systolic and Diastolic)

SECONDARY OUTCOMES:
Blood Lipid Profile | Pre-treatment and 12 weeks post-treatment
  Blood lipid profile including total cholesterol, LDL-cholesterol, HDL-cholesterol and triacylglycerides

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to other researchers. Group data could be asked by demand

REFERENCES:
- [Result] Serrano JCE, Castro-Boque E, Garcia-Carrasco A, Moran-Valero MI, Gonzalez-Hedstrom D, Bermudez-Lopez M, Valdivielso JM, Espinel AE, Portero-Otin M. Antihypertensive Effects of an Optimized Aged Garlic Extract in Subjects with Grade I Hypertension and Antihypertensive Drug Therapy: A Randomized, Triple-Blind Controlled Trial. Nutrients. 2023 Aug 23;15(17):3691. doi: 10.3390/nu15173691. PMID 37686723